CLINICAL TRIAL: NCT05638594
Title: A Randomized Controlled, Open-label, Multicenter Clinical Study of Pyrotinib Maleate Combined With Trastuzumab,Dalpiciclib, and Letrozole Versus Trastuzumab Combined With Pertuzumab, Docetaxel, and Carboplatin as Neoadjuvant Therapy for Stage II-III HR +/HER2 + Breast Cancer
Brief Title: Pyrotinib Combined With Trastuzumab, Dalpiciclib, Letrozole Versus TCbHP (Trastuzumab Plus Pertuzumab With Docetaxel and Carboplatin) as Neoadjuvant Treatment in HR +/HER2 + Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN-09
Record Dates: First submitted 2022-11-24; First posted 2022-12-06 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; dalpiciclib; Letrozole; pertuzumab; Docetaxel; Carboplatin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyrotinib +trastuzumab+dalpiciclib+letrozole (Experimental): Every 4 weeks for 5 cycles. Cumulative 20 weeks of treatment. Premenopausal patients need to receive ovarian function suppression
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Dalpiciclib; Drug: Letrozole; Drug: Gonadotropin-releasing hormone agonist
- Trastuzumab + pertuzumab + docetaxel + carboplatin (Active Comparator): Every 3 weeks for 6 cycles. Cumulative 18 weeks of treatment
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Pyrotinib — 320mg, qd
  Arms: Pyrotinib +trastuzumab+dalpiciclib+letrozole
Drug: Trastuzumab — 8 mg/kg first dose, then 6 mg/kg，q3w
  Other Names: Herceptin
Drug: Dalpiciclib — 125mg , qd，d1-21, q4w
  Arms: Pyrotinib +trastuzumab+dalpiciclib+letrozole
Drug: Letrozole — 2.5mg，qd
  Arms: Pyrotinib +trastuzumab+dalpiciclib+letrozole
Drug: Pertuzumab — 840 mg first dose, then 420 mg, q3w
  Other Names: Perjeta
  Arms: Trastuzumab + pertuzumab + docetaxel + carboplatin
Drug: Docetaxel — 75 mg/m2, q3w
  Arms: Trastuzumab + pertuzumab + docetaxel + carboplatin
Drug: Carboplatin — AUC 6, q3w
  Arms: Trastuzumab + pertuzumab + docetaxel + carboplatin
Drug: Gonadotropin-releasing hormone agonist — Every 4 weeks for 5 cycles, premenopausal patients only
  Arms: Pyrotinib +trastuzumab+dalpiciclib+letrozole

SUMMARY:
This is an investigator-initiated randomized controlled, open-label, multicenter, prospective Phase 2 clinical study. Patients with stage II-III HR +/HER2 + breast cancer were randomly divided into two groups at a ratio of 1:1. The experimental group received pyrotinib combined with trastuzumab, dalpiciclib and letrozole; the control group received trastuzumab combined with pertuzumab, docetaxel and carboplatin. The main study objective was to evaluate the efficacy and safety of neoadjuvant therapy for HR +/HER2 + breast cancer in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 -75 ;
2. Willing to receive LHRH agonist therapy (premenopausal patients only);
3. All patients were histopathologically confirmed to be estrogen receptor (ER) -positive and HER2-positive.
4. Treatment-naïve stage II-III patients with tumor stage meeting AJCC version 8 criteria;
5. ECOG score 0-1;
6. Organ function level must meet the following requirements:

(1) bone marrow function • ANC ≥ 1.5 x 109/L ; • PLT ≥ 100 × 109/L • Hb ≥ 90 g/L ; (2) hepatic and renal function • TBIL ≤ 1.5 × ULN; • AL and AST ≤ 3 × ULN (ALT and AST ≤ 5 × ULN in patients with liver metastases); • BUN and Cr ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min; (Cockcroft-Gault formula) (3) Echocardiography: LVEF ≥ 50%; (4) 12-lead ECG: QT interval ≤ 480 ms; 7. Able to undergo needle biopsy; 8. Voluntarily join this study to sign informed consent, have good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

1. Received any form of anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
2. Received any other anti-tumor therapy at the same time;
3. Bilateral breast cancer, inflammatory breast cancer or occult breast cancer;
4. Stage IV breast cancer;
5. Breast cancer without histopathological diagnosis;
6. Other malignant tumors in the past 5 years, except cured cutaneous basal cell carcinoma and cervical carcinoma in situ;
7. Severe heart, liver and kidney and other vital organ dysfunction;
8. Inability to swallow, chronic diarrhea and intestinal obstruction, there are a variety of factors affecting drug administration and absorption;
9. Participated in other drug clinical trials within 4 weeks before enrollment;
10. Known history of hypersensitivity to the drug components of this protocol; history of immunodeficiency, including positive HIV test, HCV, active viral hepatitis B or other acquired, congenital immunodeficiency diseases, or history of organ transplantation;
11. Had any cardiac disease, including: (1) cardiac arrhythmia requiring medication or clinically significant; (2) myocardial infarction; (3) heart failure; (4) any other cardiac disease judged by the investigator to be inappropriate for participation in this trial;
12. Female patients who are pregnant or lactating, female patients of childbearing potential with a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
13. According to the investigator 's judgment, there are concomitant diseases that seriously jeopardize the patient' s safety or affect the patient 's completion of the study (including but not limited to uncontrolled severe hypertension, severe diabetes, active infection, etc.);
14. Had a documented history of neurological or psychiatric disorders, including epilepsy or dementia.Any other condition that, in the opinion of the investigator, would make the patient inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate (tpCR: ypT0-is/ypN0) | 3 years
  Proportion of patients without any residual invasive cancer in pathological assessment of hematoxylin and eosin-stained resected breast cancer samples and all ipsilateral lymph node samples following completion of neoadjuvant therapy and surgery

SECONDARY OUTCOMES:
Best overall response | 3 years
  Proportion of patients with tumor response at any time during the study
Breast Pathologic Complete Response Rate (bpCR: ypT0-is) | 3 years
  Proportion of patients without any residual invasive carcinoma in pathological assessment of hematoxylin and eosin stained resected breast cancer samples following completion of neoadjuvant therapy and surgery.
Residual cancer burden (RCB) | 3 years
  RCB score is obtained according to pathological evaluation after completion of neoadjuvant treatment and surgery

OTHER OUTCOMES:
Disease-free survival (DFS) | 6 years
  It refers to the length of time from the start of medication after enrollment to the death of the patient because of the recurrence, distant metastasis of the disease, invasive contralateral breast cancer, or any other cause
Overall survival (OS) | 10 years
  It refers to the length of time from the start of treatment to the death of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huo S, Xue J, Wang S, Shan H, Chen G, Niu N, Wang Y, Qiu F, Zhao Y, Xing F, Zheng X, Tu W, Li K, Zhao H, Tang M, Xu Q, Liu C, Zhao Y, Jiang X, Pang Z, Zhang K, Zhang D, Chen ZS, Liu C. A pilot trial of neoadjuvant pyrotinib plus trastuzumab, dalpiciclib, and letrozole for triple-positive breast cancer. MedComm (2020). 2024 Mar 10;5(3):e505. doi: 10.1002/mco2.505. eCollection 2024 Mar. PMID 38469548